CLINICAL TRIAL: NCT04226521
Title: Extracorporeal Photopheresis for the Prevention of Early Cardiac Allograft Vasculopathy Detected by Optical Coherence Tomography
Brief Title: Extracorporeal Photopheresis and Early Cardiac Graft Vasculopathy
Acronym: ECP-OCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bosko Skoric (Other)
Collaborators: University of Zagreb (Other)
Responsible Party: Sponsor-Investigator, Bosko Skoric, Asst. prof., University of Zagreb
Organization: University of Zagreb (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ECP-OCT2019
Record Dates: First submitted 2019-09-29; First posted 2020-01-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Cardiac Allograft Vasculopathy; Heart Transplant Rejection
Keywords: Heart transplant; vasculopathy; extracorporeal photopheresis; prevention; optical coherence tomography
MeSH Terms: conditions — Vascular Diseases

STUDY DESIGN:
Intervention Model Description: Patients are randomized after heart transplant into two groups. Those randomized for extracorporeal photopheresis undergo 10 procedures during first year, in addition to standard follow-up. Patients in the control group are treated and followed-up according to standard protocol of our transplant center.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Photopheresis (Experimental): Patients who sign informed consent form undergo prophylactic extracorporeal photopheresis after heart transplant according to predetermined protocol
  Interventions: Procedure: Extracoropreal photopheresis
- No prophylactic photopheresis (No Intervention): Standard post-transplant protocol without prophylactic extracorporeal photopheresis

INTERVENTIONS:
Procedure: Extracoropreal photopheresis — Patients who sign informed consent form undergo prophylactic extracorporeal photopheresis after heart transplant according to predetermined protocol
  Arms: Photopheresis

SUMMARY:
Heart transplantation is a golden standard for the treatment of terminal heart failure. The major cause of death in late posttransplant period is cardiac allograft vasculopathy (CAV). This posttransplant complication develops slowly over several years, and when diagnosed either by conventional coronary angiography or due to graft failure, it is often too advanced and difficult to treat since it is diffuse coronary artery disease.

Therefore, early prevention of CAV is a subject of major interest in the transplant cardiology. Since CAV is associated with immune factors, immunomodulatory therapeutic options, like extracorporeal photopheresis are lately being investigated.

Unlike conventional coronary angiography, optical coherence tomography (OCT) is able to detect the development of CAV in the earliest phase, i.e. even in the first post-transplant year.

In our study, we plan to investigate the prophylactic effect of extracorporeal photopheresis in the early development of cardiac graft vasculopathy detected by OCT.

DETAILED DESCRIPTION:
Introduction

Heart transplant is golden standard in the treatment of terminal heart failure. Although patients' survival improved due to new advanced surgical techniques and the use of modern immunosuppressants, the posttransplant period of these patients is still fraught with complications and associated with reduced life expectancy compared to healthy individuals. Morbidity and mortality in the early post-transplant period are mainly associated with infections, acute graft rejection, multiorgan failure, and unspecified graft failure. In the late posttransplant period, the main cause of death is cardiac allograft vasculopathy (CAV). It should be emphasized that 30% of patients after 5 years and 50% after 10 years have angiographic changes in coronary arteries. Unlike atherosclerosis in the native heart that is typically focal, noncircumferential and usually localized in proximal segments of coronary arteries, CAV is a diffuse disease with concentric intimal hyperplasia and thickening of microvasculature media. It is a multifactorial disease caused by the immune, but also other non-immune factors: cellular and humoral (antibody-mediated) graft rejection, donor-specific anti-HLA antibodies, CMV infection, and hypercholesterolemia. The pathophysiology of immune-mediated development of CAV is based on T-cell and vascular endothelial interaction. According to the previously known association between graft rejection and development of coronary vasculopathy, routine clinical follow-up of transplanted patients includes regular myocardial biopsies with pathohistological analysis for cellular and humoral rejection.

Although CAV sometimes develops rapidly, it is usually slowly progressive disease associated with the development of chronic humoral graft rejection. Since symptoms and signs of CAV are usually absent or atypical (due to afferent and efferent graft denervation), early diagnosis is extremely important. For that reason, according to current recommendations of International Society for Heart and Lung Transplantation (ISHLT), regular periodic coronary angiographies are being performed. Nowadays, modern transplant centers, besides classical coronary angiography, perform intravascular ultrasound (IVUS) for coronary artery imaging. It provides a measurement of intimal thickness and today it is the gold standard in early detection of vasculopathy. However, due to the better spatial resolution of coronary artery layers, especially the intimal layer, in comparison to IVUS, optical coherence tomography (OCT) is started to use more often in the detection of CAV.

Despite many efforts, there are still no effective measures for CAV prevention. Out of all examined options, statin therapy and use of mTOR inhibitors as a part of the immunosuppressive regimen is providing best, but still not effective enough. Since the development of CAV is associated with various immune factors, immunomodulatory therapeutic options are being investigated. One of those options is extracorporeal photopheresis. It is an immunoregulatory method that divides patients' peripheral blood into two fractions: leukocyte-rich and leukocyte-poor fraction. The first fraction is immediately returned in circulation, and another one is exposed to UVA irradiation to achieve the immunomodulatory effect, i.e. increase in regulatory T-cell activity. This reduces rejection and graft vasculopathy as a result of an excessive immune response to the transplanted organ. The positive effect of this therapeutic method on CAV development was confirmed in one small study where pathomorphological changes of coronary arteries were detected using IVUS. Moreover, maintenance immunosuppressive therapy in study patients included a combination of cyclosporin and azathioprine, inferior to contemporary immunosuppressive combinations.

Hypothesis Extracorporeal photopheresis, along with other standard methods of treatment after heart transplantation significantly reduces the development of cardiac allograft vasculopathy as detected with optical coherence tomography.

Materials and methods:

This is a controlled prospective study of de novo heart transplant patients followed at the the Department for intensive care unit, arrhytmias and transplantation cardiology at University Hospital Center Zagreb. We plan to enroll 25 consecutive patients after heart transplant after signing an informed consent form. All patients will be treated with standard immunosuppressive protocol and have a standard follow-up with regular biopsies. The number of patients (12-13) determined by chance will receive additional treatment with extracorporeal photopheresis (ECP) according to a predetermined protocol. During the first post-transplant year, these patients will undergo 10 ECP treatments, each pair of treatment given on two consecutive days. Complete blood count, electrolytes and coagulation parameters are performed prior to the procedure. Since psoralen application can cause photosensitivity, patients are advised to avoid sun exposure for 24 hours. The procedure will be performed in the Department for transfusion and transplantation biology at University Hospital Center Zagreb.

All patients included in the study will undergo two coronary angiographies with OCT imaging - the initial within the first three months after heart transplantation, and the second 12 months after heart transplantation. Ilumien Optis System platform with Dragonfly Optis Imaging catheter will be used to acquire high-resolution images. OCT images acquired at basal and control will be used for statistical analysis of ECP effect on the development of cardiac allograft vasculopathy. OCT acquisition will be performed in all three major coronary arteries. The analysis will be performed in a blinded fashion. For quantification of intimal tissue hyperplasia, we will measure maximal and median intimal thickness, maximal and mean intima area, as well as volumetric indices including intimal volume, plaque volume, and plaque index. These parameters will be normalized to measured segment length. Qualitative intimal tissue analysis will be performed as well. All plaques in the acquired segments will be characterized and sized according to luminal presentation and mapped for serial assessment.

During the study, we will collect patients' medical history data, anthropometric measurements, and laboratory tests results. According to the standard protocol of myocardial biopsies and pathological analysis, results regarding graft rejection will be used in the comparative analysis of photopheresis efficacy.

ELIGIBILITY:
Inclusion Criteria:

* age >18 and <65
* primary orthotopic heart transplant
* early photopheresis
* adequate intravenous approach
* signed informed consent

Exclusion Criteria:

* aphakia
* psoralen hypersensitivity
* active retinal disease - photosensitive diseases
* splenectomy
* L <2000; Hb <70 g/L
* coagulopathy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2023-10-17 (Actual); Study Completion 2023-10-17 (Actual)

PRIMARY OUTCOMES:
Prevention of cardiac allograft vasculopathy detected by optical coherence tomography | One year
  It will be measured as the mean change in maximal intimal thickness (mm) between matched slices and the mean change in intimal volume (mm3) between matched coronary segments from baseline to month 12. Intima-to-media border will be identified as sharp line between first bright layer (intima) and first dark layer (media) of vessel wall. OCT will be performed during the patient's angiogram at baseline (1-3 months after transplantation) and again at one year after transplantation. An attempt will be made to get OCT image of all three coronary arteries. Two independent experienced angiographers, who will be blinded to clinical data, will review the baseline and follow-up image acquisition sequences to accurately match the coronary segments. We will compare the mean change of maximal intimal thickness (mm) and/or the mean change of intimal volume (mm3) between patients who underwent extracorporeal photopheresis (ECP) to those who did not undergo ECP.

SECONDARY OUTCOMES:
Number of patients with angiographically detected coronary artery disease | 1 year
  Angiographically detected CAV is defined as any new luminal irregularity or new stenosis ≥50% on control coronary angiography at 12 months interval.
  We will compare the incidence of angiographically detected transplant vasculopathy defined as newly occurring angiographic luminal irregularities or ≥50% stenosis between patients who underwent extracorporeal photopheresis (ECP) to those who did not undergo extracorporeal photopheresis (ECP).
Number of patients with acute cellular rejection | 1 year
  Patients will be monitored for acute rejection by routine surveillance endomyocardial biopsy at 1, 2, 4, 6, 9 and 12 months after heart transplantation. Graft rejection will be as an acute cellular rejection with histopathology grade ≥1B according to the 1990 International Society of Heart and Lung Transplantation classification and ≥2R according to the 2004 R grading system. For patients with multiple episodes of rejection, the time to the first event will be counted as the censored outcome. A 1-year cumulative total rejection score (TRS) will be assigned as grade 0=0, grade 1A=0.5, grade 1B=1, grade 2=1.5, grade 3A=2, grade 3B=2.5, grade 4=3, or as grade 0R=0, grade 1R = 1, grade 2R=2, grade 3R=3, and normalized by dividing the cumulative scores with the total number of biopsies performed during the 1-year period. We will compare the incidence of acute cellular rejection between patients who underwent ECP to those who did not undergo ECP.
Number of patients with antibody-mediated rejection | 1 year
  Patients will be monitored for antibody-mediated rejection (AMR) by routine surveillance endomyocardial biopsy at 1, 6 and 12 months within the first year after heart transplantation. It will be defined as either positive immunopathologic finding (the presence of C4d deposition in capillaries in the fresh-frozen biopsy sample), positive histopathologic finding or both.
  We will compare the incidence of antibody-mediated rejection between patients who underwent extracorporeal photopheresis (ECP) to those who did not undergo extracorporeal photopheresis (ECP).
Number of patients with positive donor specific antibodies | 1 year
  Patients will be monitored for de novo donor specific antibodies (DSA) by routine laboratory surveillance using Luminex assay at 1, 6 and 12 months within the first year after heart transplantation. Positive DSA will be defined as donor-specific antibody with mean fluorescence intensity (MFI) ≥ 2000.
  We will compare the incidence of positive de novo donor specific antibodies between patients who underwent extracorporeal photopheresis (ECP) to those who did not undergo extracorporeal photopheresis (ECP).
Left ventricular function expressed as ejection fraction (%) and plasma levels of NT-proBNP | 1 year
  Left ventricular systolic function will be assessed by echocardiography and expressed as ejection fraction (%), as well as plasma levels of N-terminal prohormone of brain natriuretic peptide (NT-proBNP) (ng/L) measured at month 12.
  We will compare left ventricular ejection fraction and NT-proBNP plasma concentration at month 12 between patients who underwent extracorporeal photopheresis (ECP) to those who did not undergo extracorporeal photopheresis (ECP).
Levels of T-lymphocyte subsets, B-lymphocytes, and NK cells in peripheral blood evaluated by the flow cytometry technique | 1 year
  Peripheral blood samples will be taken just before transplantation, and then before 6th and 9th ECP cycle. Sample will be taken before leukapheresis and analyzed for WBC, hematocrit, mononuclear cells (MNC), and platelet counts. Number of T-lymphocyte subsets (CD3+, CD3+4+, CD3+8+, CD4+8+ ratio) B-lymphocytes (CD 19+), and NK cells (CD56+) in patient's peripheral blood will be taken according to schedule. The levels of T, B lymhocytes and NK cells will be evaluated by the flow cytometry technique (Becton Dickinson, Facs Calibur, USA). The values of lymphocyte subsets will be expressed as percentages and absolute counts (cells/μl).
Number of patients with adverse events - safety assesments | 1 year
  Safety will be assessed by the number of patients with adverse events including: death, all infections (pneumonia, CMV viremia/infection, urinary tract infection, wound infection, sepsis…), CMV viremia/infection, indwelling venous access catheters related bacteremia, indwelling venous access catheters related thrombosis. CMV will be documented as infection (viremia) and disease (viremia with clinical symptoms and signs).

CONTACTS AND LOCATIONS:
Overall Officials: Boško Skorić, Principal Investigator — UHC Zagreb
Locations (1):
- UHC Zagreb, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF
Time Frame: The data will be available in 2 years for time frame of 5 years